CLINICAL TRIAL: NCT03754998
Title: Community Interventions to Improve Iron and Iodine Status in Mother and Child Dyads in Northern Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Won O. Song, Professor, Michigan State University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: WSong
Record Dates: First submitted 2018-11-14; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Iron Deficiency (ID); General Anemia; Iron Deficiency Anemia (IDA)
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency

STUDY DESIGN:
Intervention Model Description: Quasi experimental
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): The participating dyads in intervention communities were invited to consume veo soup/meal (HSM) three times a week and provided weekly supply of iodized salt (450 g) for the household usage as well as being engaged in dry season container gardening. The veo soup/meal is a local Ghanaian soup/meal mainly made of Hibiscus Sabdarifa leaves. It is a soup when prepared a bit watery and consumed with 'tou zaafi' (millet or corn based cooked paste). It is also a meal when prepared thick and eaten by itself. The Hibiscus Sabdariffa leaves meal (HSM) used in the present study was made of 18 kg Hibiscus Sabdariffa leaves, 8 kg groundnut, 1.1 kg dawadawa (fermented African locust beans), 3 kg dried fish plus 0.045 kg iodized salt, cooked with about 23 L (23 kg) water to yield 52.5 kg HSM. In each community, groups of ten women took turns to share the cooking activities, washing of bowls, and making water available for cooking. No treatment provided in our control communities.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — The participating dyads in intervention communities were invited to consume veo soup/meal (HSM) three times a week and provided weekly supply of iodized salt (450 g) for the household usage as well as being engaged in dry season container gardening. The veo soup/meal is a local Ghanaian soup/meal mainly made of Hibiscus Sabdarifa leaves. It is a soup when prepared a bit watery and consumed with 'tou zaafi' (millet or corn based cooked paste). It is also a meal when prepared thick and eaten by itself. The Hibiscus Sabdariffa leaves meal (HSM) used in the present study was made of 18 kg Hibiscus Sabdariffa leaves, 8 kg groundnut, 1.1 kg dawadawa (fermented African locust beans), 3 kg dried fish plus 0.045 kg iodized salt, cooked with about 23 L (23 kg) water to yield 52.5 kg HSM. In each community, groups of ten women took turns to share the cooking activities, washing of bowls, and making water available for cooking. No treatment provided in our control communities.

SUMMARY:
BACKGROUND Ghana has reduced food insecurity prevalence by 49.2% in two decades. However, prevalence of malnutrition especially stunting (in <children5yr) has not matched the changes in food security levels. Of several key nutritional factors that lead to stunting, nutritional status of such trace minerals as iodine, iron and zinc has not been studied. Nutritional inadequacy of these trace minerals may be detected by estimation of dietary intake, and time-consuming and costly biochemical measurements of respective biomarkers. Since there is no means to estimate dietary intake of the trace minerals in Ghana, due to incomplete food composition data of the nutrients, identifying validated non-invasive, dietary approaches to predict the biomarker status of these trace minerals are critical in counteracting the challenges surrounding the persistent stunting due to micronutrient deficiencies in Ghana. Additionally, exploring alternative approaches to providing access to foods rich in trace minerals at household level is crucial.

STUDY AIMS AND HYPOTHESIS The ultimate goal of this research is to increase knowledge base on improving trace mineral status in mother-child (6-23 mo) dyads through a sustainable community-based interventions in northern Ghana. Investigators will begin with iron and iodine that impair mothers and young children's growth and cognitive development most with three aims: 1) to develop dietary screening tools that are validated by biomarkers for early detection of deficiencies, 2) to determine efficacy (dose responses) of feeding indigenous nutrient-rich meals in preventing deficiencies and improving iron and iodine status, and 3) to demonstrate sustainable and scalable improvement of food systems through a container gardening project for iron-rich Hibiscus sabdarifa for consumption and income by empowering women during the dry/lean season in northern Ghana.

• Aims 1: To develop dietary screening tools that are validated by biomarkers for early detection of deficiencies among children 6-23 months and their mothers H1.1: Dietary diversity score can predict iron deficiency among children 6-23 months and their mothers.

H1.2: Dietary diversity score can predict iodine status deficiency among children 6-23 months and their mothers.

* Aims 2: Indigenous nutrient-rich meals of hibiscus sabdarifa improves iron and iodine status of dyads H2.1: Indigenous nutrient-rich meals of hibiscus sabdarifa improves iron status of dyads H2.2: Indigenous nutrient-rich meals of hibiscus sabdarifa improves iodine status of dyads
* Aims 3: to demonstrate that container gardening can provide sustainable and scalable improvement of food systems for iron-rich Hibiscus sabdarifa for consumption and income during the dry/lean season in northern Ghana H3.1: Container gardening can provide adequate amounts of vegetables for mother and child dyad during the dry season H3.2: Container gardening can provide adequate income to purchase iodized salt and Amani for mother and child dyad during the dry season

SIGNIFICANCE This project addresses the gap in our knowledge and practices pertaining to serious and persisting trace mineral deficiencies that result in stunting and cognitive impairment in northern Ghana. Early detection of iron and iodine deficiencies with validated non-invasive dietary screening tools (aim 1), effective indigenous nutrient-rich meal-based programs (aim 2) and sustainable/scalable and women-led community-based food-system changing agricultural project (aim 3) are expected to be the most creative approach to counteract iron and iodine deficiencies in northern Ghana. This project will utilize science and education to change practices, environments and policies to reduce the prevalence of trace mineral deficiencies at the local, regional, national and global levels.

ELIGIBILITY:
Inclusion Criteria:

* Be a woman (15-49 y) and having a child (6 - 23 months)
* Live in research settings for the entire research duration (May 2016 - September 2017)
* Live in selected communities in the Kassena Nankana West and Builsa North Districts of the Upper East Region of Ghana
* Selected districts should be among the top five food insecure districts
* Households in selected communities should have access to water throughout the dry season without shortages
* Selected communities should have sizeable number of children (6 - 23 months old) for a good sampling frame

Exclusion Criteria:

Not meeting the inclusion criteria

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 239 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Iron Deficiency (ID) | 12 weeks
  ID measured using serum transferrin receptor (Stfr). Cut off for ID (women - stfr>4.40ug/l, children - stfr>2.85ug/l).
General Anemia | 12 weeks
  General anemia measured using hemoglobin levels (Hb). Cut off for General anemia (women - Hb<12g/dl, children - Hb<11g/dl)
Iron Deficiency Anemia (IDA) | 12 weeks
  IDA is measured by concurrent presence of general anemia (women - Hb<12g/dl, children - Hb<11g/dl) and ID (women-stfr>4.40ug/l, children - stfr>2.85ug/l).
Iodine status of participants | 12 weeks
  Iodine status will be measured by urinary iodine concentration (ug/l)
Hibiscus Sabdariffa produced/harvested from container gardening | 15 weeks
  Quantity of Hibiscus Sabdariffa leaves (kg) per container
Income generated form container gardening | 15 weeks
  Income (cedis) generated from cabbage produced per container

CONTACTS AND LOCATIONS:
Overall Officials: Clement Professor Won Song, Study Chair — Michigan State University; Clement Kubuga, Principal Investigator — University for Development Studies - Ghana
Locations (1):
- Builsa North and Kessena Nankana West Districts, Bolgatanga, Upper East Region, Ghana